CLINICAL TRIAL: NCT05557344
Title: Oral Versus Intravenous Acetaminophen for the Treatment of Pain Secondary to Long Bone Fracture Requiring Surgery in Children
Brief Title: Oral vs IV Acetaminophen for Long-bone Fracture in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Niina Kleiber (Other)
Responsible Party: Sponsor-Investigator, Dr. Niina Kleiber, Paediatrician and Clinical Pharmacologist, St. Justine's Hospital
Organization: St. Justine's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Acetaminophen IV vs PO
Record Dates: First submitted 2022-08-24; First posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Pain
Keywords: pain; analgesics; pediatrics; acetaminophen; orthopedics; pharmacokinetics
MeSH Terms: conditions — Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral acetaminophen arm (Active Comparator): they will receive oral acetaminophen, placebo (saline) IV
  Interventions: Drug: Acetaminophen
- IV acetaminophen arm (Active Comparator): they will receive IV acetaminophen, placebo oral
  Interventions: Drug: Acetaminophen IV

INTERVENTIONS:
Drug: Acetaminophen IV — An IV infusion of 15mg/kg of acetaminophen (PrACETAMINOPHEN INJECTION, AVIR Pharma Inc.) (maximum single dose:1g) will be administered regularly every 6h as a 15-minute intravenous infusion. At the same time, an oral placebo with similar appearance as the corresponding acetaminophen oral solution will be administered.
  Arms: IV acetaminophen arm
Drug: Acetaminophen — A liquid oral acetaminophen suspension will be administered regularly every 6h at a dose of 15mg/kg (maximum single dose: 1g). An IV infusion of NaCl 0.9% corresponding to the volume of IV acetaminophen will be administered as a 15-minute intravenous infusion at the same time as the oral dose. PrACETAMINOPHEN INJECTION ® is a clear and colorless liquid undistinguishable from NaCl 0.9%.
  Arms: Oral acetaminophen arm

SUMMARY:
Intravenous (IV) acetaminophen entered the Canadian market recently and children with acute pain following a trauma are ideal candidates for the IV formulation as it may improve analgesia and consequently decrease the amount of opioids needed to achieve pain control. Due to the limited data on bioavailability, adverse effect profile and efficacy of IV versus oral acetaminophen, it is of paramount importance to generate evidence-based data to guide clinicians with a rational choice of route of administration of acetaminophen.

Therefore, we propose a pilot study to inform a future large randomized controlled trial (RCT) to compare pharmacokinetics, feasibility, preliminary effects and side effects profile of oral versus IV acetaminophen in children admitted for surgical fixation of a long-bone fracture.

DETAILED DESCRIPTION:
Patients admitted for a long-bone fracture needing surgical fixation are generally initially treated with intranasal and/or IV opioids in association to oral acetaminophen and ibuprofen. Following surgery they are treated with a combination of morphine and acetaminophen. To address the issue of opioid epidemics, the Pediatric Orthopaedic Society of North America recommends reduction of their prescription as much as possible by promoting, among others, use of multimodal analgesia after surgery. The current proposal aims to improve post-operative pain control in children following a surgical fixation of a long-bone fracture and decrease the use of opioids through better co-analgesia. As such, this study aims to assess the pharmacokinetics (PK) and the efficacy of oral versus IV formulations of acetaminophen after surgery for long bone fractures in children.

ELIGIBILITY:
Inclusion Criteria:

* Likely to undergo surgery for a long-bone fracture
* Aged between 2-18 years (IV acetaminophen is approved for children ≥2 years)
* IV line per standard of care

Exclusion Criteria:

* Contraindication to oral drug administration
* Patients unable to take oral solution
* Known hypersensitivity or allergy to acetaminophen or any of the excipients in the IV or oral formulation
* Use of any medication known to interact with acetaminophen including, but not restricted to phenytoin and carbamazepine (1)
* Pregnancy
* Known Hepatic insufficiency or hepatic disease
* Known or diagnosed severe renal failure
* Multiple trauma (more than two long bone fractures)
* Hemodynamic or respiratory compromise
* Altered level of consciousness (Glasgow coma scale <15)

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain scores | During 24h (starting with the first dose of study drug)
  Pain scores within the first 24 hours following initiation of study drug, using the scales Face, Legs, Activity, Cry, Consolability (FLACC, 0-2 per item for a total of 10, 10 being the worst pain) and verbal numerical rating (VNR, 0-10, 10 being the worst pain).
Difference in quantity of rescue opioids | During 24h (starting with the first dose of study drug)
  Quantity of rescue opioids (morphine equivalent in mg/kg) within the first 24 hours following initiation of study drug

SECONDARY OUTCOMES:
Adverse events | During 24h (starting with the first dose of study drug)
  Any other adverse effect whether or not attributed to the study drug will be carefully recorded. Opioid-related adverse effects will be recorded (pruritus, time to first bowel movement, nausea (self-reported), vomiting, days of bladder catheterization, oxygen supplementation, episodes of respiratory depression (< 10/min in children older than 5 years), use of diphenhydramine, naloxone, antiemetics, laxatives).
Determination of oral bioavailability | During 24 hours after the first dose of study drug
  Blood level of acetaminophen will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Niina Kleiber, MD PhD, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ulrich M, Chamberland M, Bertoldi C, Garcia-Bournissen F, Kleiber N. Newly approved IV acetaminophen in Canada: Switching from oral to IV acetaminophen. Is IV worth the price difference? A systematic review. Paediatr Child Health. 2021 Mar 13;26(6):337-343. doi: 10.1093/pch/pxaa137. eCollection 2021 Oct. PMID 34676011